CLINICAL TRIAL: NCT05382559
Title: A Phase 1 Study of ASP3082 in Participants With Locally Advanced or Metastatic Solid Tumor Malignancies With KRAS G12D Mutation
Brief Title: A Study of ASP3082 in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3082-CL-0101; jRCT2031220738 (Registry Identifier: jRCT); CTR20250465 (Registry Identifier: chinaDrugTrials.org.cn); 2022-501590-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; Cancer; Malignancy; Metastasis; Pharmacokinetics; ASP3082; KRAS G12D; NSCLC; CRC; PDAC
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Leucovorin; Fluorouracil; Irinotecan; Taxes; Gemcitabine; Docetaxel; pembrolizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- ASP3082 Dose Escalation (Monotherapy Part 1) (Experimental): Participants will receive ASP3082 in a 21-day cycle.
  Interventions: Drug: ASP3082
- ASP3082 Dose Expansion (Monotherapy Part 2) (Experimental): Participants will receive ASP3082 with dose level(s) selected from dose escalation (part 1) in a 21-day cycle.
  Interventions: Drug: ASP3082
- ASP3082 + Cetuximab Dose Escalation (Combination Therapy Part 1) (Experimental): Participants will receive ASP3082 in a 21-day cycle. Cetuximab will be administered weekly.
  Interventions: Drug: ASP3082; Drug: Cetuximab
- ASP3082 + Cetuximab Dose Expansion (Combination Therapy Part 2) (Experimental): Participants will receive ASP3082 or ASP3082 + Cetuximab with dose level(s) selected from dose escalation (part 1) in a 21-day cycle. Cetuximab will be administered weekly.
  Interventions: Drug: ASP3082; Drug: Cetuximab
- ASP3082 China Safety Cohort (Experimental): Participants will receive ASP3082 with dose level selected from dose escalation (Monotherapy part 1) in a 21-day cycle.
  Interventions: Drug: ASP3082
- Treatment naive PDAC cohort ASP3082 + FOLFIRINOX (Experimental): Upon completion of dose escalation (part 1), participants with KRAS G12D mutant will receive ASP3082 in combination with FOLFIRINOX (leucovorin [LV]/fluorouracil [5-FU]/irinotecan/oxaliplatin) with dose level(s) selected from dose escalation (part 1) in a 28-day cycle.
  Interventions: Drug: ASP3082; Drug: Leucovorin; Drug: Oxaplatin; Drug: Fluorouracil; Drug: Irinotecan
- Treatment naive PDAC cohort ASP3082 + Nab-Paclitaxel + Gemcitabine (Experimental): Upon completion of dose escalation (part 1), participants with KRAS G12D mutant will receive ASP3082 in combination with Nab-P + GEM (nanoparticle albumin-bound-paclitaxel plus gemcitabine) with dose level(s) selected from dose escalation (part 1) in a 28-day cycle.
  Interventions: Drug: ASP3082; Drug: Nanoparticle albumin-bound-paclitaxel; Drug: Gemcitabine
- ASP3082 + Docetaxel - NSCLC (Experimental): Participants with KRAS G12D mutant will receive ASP3082 in combination with docetaxel in a 21-day cycle.
  Interventions: Drug: ASP3082; Drug: Docetaxel
- ASP3082 + Pembrolizumab - NSCLC (Experimental): Participants with KRAS G12D mutant will receive ASP3082 in combination with pembrolizumab in a 21-day cycle.
  Interventions: Drug: ASP3082; Drug: Pembrolizumab
- ASP3082 + (Cisplatin or Carboplatin) and Pemetrexed +/- Pembrolizumab - NSCLC (Experimental): Participants with KRAS G12D mutant will receive ASP3082 in combination with platinum-based chemotherapy (cisplatin or carboplatin) and pemetrexed, with or without pembrolizumab in a 21-day cycle.
  Interventions: Drug: ASP3082; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: ASP3082 — Intravenous Infusion
Drug: Cetuximab — Intravenous Infusion
  Arms: ASP3082 + Cetuximab Dose Escalation (Combination Therapy Part 1); ASP3082 + Cetuximab Dose Expansion (Combination Therapy Part 2)
Drug: Leucovorin — Intravenous Infusion
  Arms: Treatment naive PDAC cohort ASP3082 + FOLFIRINOX
Drug: Oxaplatin — Intravenous Infusion
  Arms: Treatment naive PDAC cohort ASP3082 + FOLFIRINOX
Drug: Fluorouracil — Intravenous Infusion
  Arms: Treatment naive PDAC cohort ASP3082 + FOLFIRINOX
Drug: Irinotecan — Intravenous Infusion
  Arms: Treatment naive PDAC cohort ASP3082 + FOLFIRINOX
Drug: Nanoparticle albumin-bound-paclitaxel — Intravenous Infusion
  Arms: Treatment naive PDAC cohort ASP3082 + Nab-Paclitaxel + Gemcitabine
Drug: Gemcitabine — Intravenous Infusion
  Arms: Treatment naive PDAC cohort ASP3082 + Nab-Paclitaxel + Gemcitabine
Drug: Docetaxel — Intravenous Infusion
  Arms: ASP3082 + Docetaxel - NSCLC
Drug: Pembrolizumab — Intravenous Infusion
  Arms: ASP3082 + (Cisplatin or Carboplatin) and Pemetrexed +/- Pembrolizumab - NSCLC; ASP3082 + Pembrolizumab - NSCLC
Drug: Cisplatin — Intravenous Infusion
  Arms: ASP3082 + (Cisplatin or Carboplatin) and Pemetrexed +/- Pembrolizumab - NSCLC
Drug: Carboplatin — Intravenous Infusion
  Arms: ASP3082 + (Cisplatin or Carboplatin) and Pemetrexed +/- Pembrolizumab - NSCLC
Drug: Pemetrexed — Intravenous Infusion
  Arms: ASP3082 + (Cisplatin or Carboplatin) and Pemetrexed +/- Pembrolizumab - NSCLC

SUMMARY:
This is an open-label study. This means that people in this study and clinic staff will know that they will receive ASP3082. The study aims to check how safe and well-tolerated ASP3082 is for people with advanced solid tumors that have a specific mutation called KRAS G12D.

This study will be in 2 parts.

In Part 1, different small groups of people will receive lower to higher doses of ASP3082 by itself, or together with cetuximab. Any medical problems will be recorded at each dose. This is done to find suitable doses of ASP3082, by itself or together with cetuximab, to use in Part 2 of the study. The first group will receive the lowest dose of ASP3082. A medical expert panel will check the results from this group and decide if the next group can receive a higher dose of ASP3082. The panel will do this for each group until all groups have received ASP3082 (by itself or together with cetuximab) or until suitable doses have been selected for Part 2.

In Part 2, ASP3082 will be given in by itself, or in combination with the other study treatments.

Study treatments will be given through a vein. This is called an infusion. Each treatment cycle is 21 or 28 days long. They will continue treatment until: they have medical problems from the treatment they can't tolerate; their cancer gets worse; they start other cancer treatment; or they ask to stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally advanced (unresectable) or metastatic solid tumor malignancy with documented Kirsten rat sarcoma viral oncogene homolog [KRAS] G12D mutation and has received prior standard therapy and the investigator does not see any further clinical benefit from continuing such targeted therapy, or is ineligible to receive or has refused standard approved therapies (no limit to the number of prior treatment regimens).
* For the ASP3082 monotherapy escalation cohorts, participants with solid tumor malignancies are allowed to be enrolled.
* For ASP3082 combination therapy with Nab-P+GEM or FOLFIRINOX: Participant must have mPDAC that has not been previously treated with chemotherapy. If a participant received (neo)adjuvant therapy, tumor recurrence or disease progression must have occurred at least 6 months after completing the last dose of the (neo)adjuvant therapy.
* Participant consents to provide tumor specimen in a tissue block or unstained serial slides or a tumor biopsy (core needle biopsy or excision) obtained after the last interventional treatment, but not more than 56 days prior to start of study intervention. Participant also consents to provide a sample for tumor biopsy during the treatment period as indicated in the study protocol. If a participant cannot provide a fresh tissue biopsy sample, the site should consult with the sponsor/study medical monitor.
* Participant has at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant has an ECOG performance status of 0, 1 or 2 for dose escalation, and 0 or 1 for dose expansion.
* Participant's last dose of prior antineoplastic therapy, including any immunotherapy, was 21 days or 5 half-lives, whichever is shorter, prior to initiation of study intervention administration.
* Participant has completed any radiotherapy (including stereotactic radiosurgery) at least 14 days prior to the start of study intervention administration. Participants must have recovered from all radiation-related toxicities, not require corticosteroids (NOTE: Physiologic replacement dose of hydrocortisone or its equivalent [defined as up to 30 mg per day of hydrocortisone, 2 mg per day of dexamethasone, or up to 10 mg per day of prednisone] is permitted), and not have active radiation pneumonitis. A 1-week washout is permitted for palliative radiation (<= 2 weeks of radiotherapy) to non-central nervous system disease.
* Participant's adverse events [AEs] (excluding alopecia) from prior therapy have improved to grade 1 or baseline within 14 days prior to start of study intervention.
* Participant has adequate organ function as indicated by protocol laboratory value parameters (If a participant has received a recent blood transfusion, the laboratory tests must be obtained >= 14 days after any blood transfusion.).
* Female participant is not pregnant, confirmed by pregnancy test and medical evaluation by interview, and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP).
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after study intervention administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 6 months after study intervention administration.
* Female participant must not donate ova starting at first dose of study intervention and throughout the study period and for 6 months after study intervention administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 3 months after study intervention administration.
* Male participant must not donate sperm during the treatment period and for 3 months after study intervention administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 3 months after study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study intervention (Participants who are currently in the follow-up period of an interventional clinical trial are allowed).

Exclusion Criteria:

* Participant has received investigational therapy within 21 days or 5 half-lives, whichever is shorter, prior to start of study intervention.
* Participant has symptomatic or untreated central nervous system (CNS) metastases. Participants with asymptomatic, treated CNS metastases are eligible.
* Participant has leptomeningeal disease as a manifestation of the current malignancy.
* Participant has a prior malignancy active (i.e., requiring treatment or intervention) within the previous 2 years, except for local malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast, which are allowed.
* Participant has a known or suspected hypersensitivity to ASP3082 or any components of the formulation used.
* Participant with active hepatitis B (including acute hepatitis B virus [HBV] or chronic HBV) or hepatitis C virus [HCV] (ribonucleic acid [RNA] detected by qualitative assay). HCV RNA testing is not required in participants with negative HCV antibody testing.
* Participant has a known history of human immunodeficiency virus [HIV] infection. No HIV testing is required unless mandated by a local health authority.
* Participant has had a myocardial infarction or unstable angina within 6 months prior to the start of study intervention, left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO) or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, obligate use of a cardiac pacemaker, or long QT syndrome.
* Participant has a corrected QT interval (single electrocardiogram [ECG]) using Fridericia's formula (QTcF) > 450 milliseconds (msec) (men) or >470 msec (women) during screening.
* Participant has received prior treatment with a specific KRAS G12D inhibitor/degrader or pan-RAS inhibitor/degrader targeting KRAS G12D. Participants who received prior treatment with a KRAS G12D inhibitor/degrader are eligible for the ASP3082 combination therapy cohort.
* Participant has an active infection requiring intravenous antibiotics within 14 days prior to study intervention.
* Participant is expected to require another form of antineoplastic therapy while on study treatment.
* Participant has any condition which makes the participant unsuitable for study participation (such as psychiatric illness/social situations that would limit compliance with study requirements).
* Participant has had major surgery within 4 weeks prior to first dose of study intervention.

For ASP3082 Combination Therapy:

* Prior discontinuation of cetuximab treatment due to toxicity or intolerance of cetuximab.
* History of interstitial lung disease requiring systemic steroid treatment. Note that a participant with resolved pulmonary infections or radiation pneumonitis is eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 21 Days
  A DLT is defined as any event meeting the DLT criteria occurring within 21 days of first dose on Cycle 1 Day 1 (C1D1), excluding toxicities clearly related to disease progression or intercurrent illness.
Number of Participants with Adverse Events (AEs) | Up to 48 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study IP, whether or not considered related to the study investigational product (IP).
  Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study IP. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants with Serious Adverse Events (SAEs) | Up to 48 months
  An SAE is defined as any untoward medical occurrence that, at any dose:
  Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and other medically important events.
Number of Participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 48 months
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with electrocardiogram (ECG) abnormalities and/or adverse events (AEs) | Up to 48 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants with vital sign abnormalities and/or adverse events (AEs) | Up to 48 months
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with physical exam abnormalities and/or adverse events | Up to 48 months
  Number of participants with potentially clinically significant physical exam values.
Number of Participants with Eastern Cooperative Oncology Group (ECOG) performance status | Up to 48 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 48 months
  ORR is defined as the proportion of participants whose best overall response is rated as complete response (CR) or partial response (PR) per RECIST v1.1.
Duration of Response (DOR) per RECIST v 1.1 | Up to 48 months
  DOR is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date of documented radiological disease progression per RECIST v1.1 or death in the absence of progression.
Disease Control Rate (DCR) per RECIST v 1.1 | Up to 48 months
  DCR is defined as the proportion of participants whose best overall response is rated as CR, PR or SD based on RECIST v1.1.
Pharmacokinetics (PK) of ASP3082 in plasma: Area under the concentration-time curve (AUC) | Up to 48 months
  AUC will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: Maximum Concentration (Cmax) | Up to 48 months
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 48 months
  Ctrough will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: Time of maximum concentration (tmax) | Up to 48 months
  tmax will be recorded from the PK plasma samples collected.
Changes in Kirsten rat sarcoma (KRAS) viral oncogene homolog G12D in tumor samples | Up to 48 months
  Changes in KRAS G12D in tumor samples will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (49):
- United States (22):
  - City of Hope National Medical Center, Duarte, California
  - UCLA Santa Monica Hematology Oncology, Santa Monica, California
  - Denver HealthONE Drug Development Unit, Denver, Colorado
  - Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida, Davis Cancer Center, Gainesville, Florida
  - Florida Cancer Specialist, Lake Mary, Florida
  - Florida Cancer Specialists & Research Institute Sarasota, Sarasota, Florida
  - University of Kansas Medical Center, Westwood, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Wisconsin Hospital, Madison, Wisconsin
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Xuhui District, Shanghai Municipality
- France (5):
  - Site FR33003, La Tronche, Grenobele
  - Site FR33002, Bordeaux
  - Site FR33001, Lyon
  - Site FR33005, Lyon
  - Site FR33004, Villejuif, Île-de-France Region
- Japan (12):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kindai University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Osaka International Cancer Institute, Osaka
- South Korea (4):
  - Site KR82002, Seongnam-si, Gyeonggi-do
  - Site KR82001, Jongno -Gu, Seoul
  - Site KR82003, Seodaemun-gu, Seoul
  - Site KR82004, Songpa-gu, Seoul
- Spain (4):
  - Site ES34001, Barcelona
  - Site ES34004, Madrid
  - Site ES34002, Málaga
  - Site ES34003, Seville

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/